CLINICAL TRIAL: NCT04580017
Title: Prognostic Accuracy of the HEART Score in Undifferentiated Chest Pain: A Multicenter Validation Study
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professeur, University of Monastir
Other Study IDs: HEART score
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Coronary Disease; Coronary Syndrome; Risk Factor, Cardiovascular; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Coronary Disease; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chest pain remains one of the most common, potentially serious presenting complaints for adults emergency department visits with approximately 7.6 million yearly visits in the united states. The priority for emergency physician is to determine whether these patients with acute chest pain have a potential life threatening underlying etiology. The great challenge is to differentiate patients presenting with acute coronary syndrome and those with other more benign conditions.

There is a global tendency for ED physician to over investigate chest pain patients , even in low-risk patients. This kind of practice leads to resource over-utilization and a huge health costs waste contrasting with no outcomes improvement.

For many years, physicians have been searching tools, ranging from specific diagnostic tests to entire strategies of evaluation, to appropriately stratify the risk in patients with chest pain in order to simultaneously prevent major adverse cardiac events and reduce unnecessary testing and hospitalizations. Many bioclinical scores have been developed, such as the TIMI score and the GRACE score.The HEART score is one of the more recently proposed model derived through a process involving expert opinion and review of medical literature. It is calculated based on admission data of medical history, EKG, age, cardiovascular risk factors and troponin levels.

The HEART score was created specifically to identify ED patients presenting with undifferentiated chest pain who were at low risk as well as patients at high risk of short-term MACE occurrence. HEART score has been widely reported to outperform the TIMI and the GRACE scores. Several scientific societies are encouraging the use of HEART score, for evaluating patients with chest pain suggestive of ACS in the ED.

The goal of our investigation is to validate HEART score as a prognostication tool among ED patients with chest pain in teaching hospitals in Tunisia.

DETAILED DESCRIPTION:
Chest pain remains one of the most common, potentially serious presenting complaints for adults emergency department visits with approximately 7.6 million yearly visits in the united states. The priority for emergency physician is to determine whether these patients with acute chest pain have a potential life threatening underlying etiology. The great challenge is to differentiate patients presenting with acute coronary syndrome and those with other more benign conditions. Obviously, medical history, clinical examination, and laboratory values may help to identify patients with true ACS. None are sufficiently accurate to be used independently. Thus, about 5% of ACS patients are inappropriately discharged annually. Therefore, there is a global tendency for ED physician to overinvestigate chest pain patients with further, often more invasive testing, even in low-risk patients. This kind of practice leads to resource overutilization and a huge health costs waste contrasting with no outcomes improvement.

For many years, physicians were searching tools, ranging from specific diagnostic tests to entire strategies of evaluation, to appropriately risk stratify patients with chest pain in order to simultaneously prevent major adverse cardiac events and reduce unnecessary testing and hospitalisations. Based on the principal that a prompt quick and accurate identification of patients who are at high and low risk of developing major adverse cardiac events is paramount, and in order to optimally allocate ED and hospital resources, many bioclinical scores have been developed. One of the most known risk scores is TIMI score, which was originally derived and validated in a population of in-patients with unstable angina and non ST elevation myocardial infarction (NSTEMI). Its main performance is to predict early occurrence of major cardiovascular events (MACE). However, TIMI score like many other specific scores gave conflicting results when applied on chest pain patients in the ED. The HEART score is one of the more recently proposed model derived through a process involving expert opinion and review of medical literature. It is calculated based on admission data of medical history, EKG, age, cardiovascular risk factors and troponin levels. The HEART score was created specifically to identify ED patients presenting with undifferentiated chest pain who were at low risk as well as patients at high risk of short-term MACE occurrence. HEART score has been widely reported to outperform the TIMI and the GRACE scores. Several scientific societies are encouraging the use of HEART score, for evaluating patients with chest pain suggestive of ACS in the ED. A recent systematic review comprehensively compared the leading clinical prediction rules for chest pain, including the TIMI, the HEART, and the GRACE scores. Among the three risk stratification tools, the HEART score was found to be the most useful for managing patients with undifferentiated chest pain who present to the ED because it is simple, easy, and quick to use and it also has been validated in several studies conducted in the ED. Additional studies providing further worldwide data about the validation of this risk score will empower emergency physicians' decision making when relying on this score in ruling in or ruling out their chest pain patients. The goal of our investigation is to validate HEART score as a prognostication tool among ED patients with chest pain in teaching hospitals in Tunisia.

ELIGIBILITY:
Inclusion Criteria:

* Any adult aged older than 30 years.
* Chief complaint of ''chest pain'', ''chest tightness'', or ''chest pressure''.

Exclusion Criteria:

* Shortness of breath without chest pain
* ST elevation myocardial infarction (STEMI)
* Patients lost to follow up
* Patients with obvious diagnosis made immediately after initial medical evaluation

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged over 30 years admitted to the ED with typical chest pain with an EKG not showing STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 4267 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Mace | 30 days
  Rate of MACE occurence including all-cause mortality, non-fatal myocardial infarction (MI), and coronary revascularisation within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira semir, MD, Principal Investigator — CHU fattouma Bourguiba Monastir
Locations (3):
- Tunisia (3):
  - Sahloul University Hospital, Hammam Sousse, Sousse Governorate
  - Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir
  - Emergency department of university hospital Farhad Hached, Sousse, Sousse